CLINICAL TRIAL: NCT04238949
Title: The Impact of Community Health Workers in Pediatric Patients With Newly Diagnosed Type 1 Diabetes - A Pilot Study
Brief Title: Community Health Workers in Pediatric Patients With Newly Diagnosed Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-016871
Record Dates: First submitted 2020-01-21; First posted 2020-01-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus; Psychosocial Problem; Compliance, Patient; Health Behavior
Keywords: Community Health Worker; Lay Worker; Community Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Patient Compliance; Health Behavior

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Diabetes Care Group (No Intervention): Patients receive standard diabetes care.
- Community Health Worker Group (Experimental): Patients are assigned a community health worker for the first year in addition to standard diabetes care. They do not receive a community health worker for the second year of the study.
  Interventions: Other: Community Health Worker added to diabetes team

INTERVENTIONS:
Other: Community Health Worker added to diabetes team — A Community Health Worker will be added to the diabetes team caring for a child with new onset type 1 diabetes for 1 year. The intervention includes social determinants of health screening and goal setting, with home visits.
  Arms: Community Health Worker Group

SUMMARY:
The primary aim of this pilot randomized controlled trial is to determine if the integration of a Community Health Worker (CHW) into the healthcare team of children with newly diagnosed type 1 diabetes is associated with an improvement in diabetes control. The secondary objectives are to determine if utilization of CHWs is also associated with improvements in psychosocial outcomes, healthcare utilization, and decreased costs.

DETAILED DESCRIPTION:
Lower socioeconomic status (SES) is associated with adverse outcomes in children with type 1 diabetes. These children have poorer glycemic control, lower quality of life, and increased healthcare utilization. Previous efforts to improve outcomes in this patient population have focused on high-cost, high-intensity educational interventions. These efforts have been ineffective in improving clinical outcomes in patients with low SES. Adverse social determinants of health (SDOH) including food insecurity, parental unemployment and housing insecurity are extremely prevalent in under-resourced patients and their families.

Community health workers (CHWs) are trained non-medical members of the community who are empowered to address adverse SDOH through home visits and connecting patients to community resources. CHWs can assist in navigating healthcare and social services systems, reducing family stress, and breaking down community barriers to positive health behavior.

Investigators hypothesize that interventions focused on addressing adverse SDOH will reduce barriers to optimal diabetes outcomes in this patient population.

At the diabetes center at The Children's Hospital of Philadelphia (CHOP), a CHW will be assigned for one year to newly diagnosed patients with type 1 diabetes with government insurance. The support provided for this year will be tailored to the patient's needs, and may include problem solving surrounding issues related to work/education, accessing healthcare/medications, engagement with the healthcare team, transportation, housing or food insecurity. Interactions with patients will be through home visits, telephone encounters, text messaging or email. Patients will be followed for a total of two years to evaluate if improvements in outcomes are sustained after the discontinuation of CHW support.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged < 17 years old
* Within 31 days of clinical diagnosis of Type 1 Diabetes (T1D)
* Government insurance at time of enrollment
* Patient lives in a zip code in Pennsylvania within a 30-minute drive of Children's Hospital of Philadelphia (CHOP) Buerger Center for Advanced Pediatric Care at time of enrollment
* Plans on completing the "Type 1 Year 1" program at CHOP, an intensive T1D education program that is standard of care for all newly diagnosed patients with T1D at CHOP
* Diabetes autoantibody positive
* English speaking caregiver and patient

Exclusion Criteria:

* Diabetes autoantibody negative
* Children in custody of the State where there is no identified caretaker who can complete study procedures
* Non English speaking primary caregiver and patient
* Medicare insurance
* Tricare insurance
* Move to a zip code greater than a 60-minute drive from CHOP Buerger Center for Advanced Pediatric Care during the course of the study
* Move to a zip code not in Pennsylvania during the course of the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 2 years
  Improvement in glycemic control, as measured by hemoglobin A1c

SECONDARY OUTCOMES:
Hospital admissions | 2 years
  Data will be extracted from the medical record of each patient to obtain information on the number of hospital admissions.
Missed outpatient appointments | 2 years
  Data will be extracted from the medical record of each patient to obtain information on the number of attended outpatient appointments.
Emergency Department utilization | 2 years
  Data will be extracted from the medical record of each patient to obtain information about the number of Emergency Department (ED) visits
Quality of life (primary care giver) | 2 years
  The primary care giver will complete the 36-item "PedsQL Health related quality of life for parents of children with chronic disease" questionnaire using a 5-point Likert rating scale to assess how their child's illness has had an impact on their quality of life. This scale ranges in score from 0 to 144, with higher scores consistent with decreased quality of life.
Primary caregiver's diabetes self-efficacy | 1.5 years
  The 17-item, "Parental self efficacy in diabetes scale" will be completed by the primary caregiver using a 5-point Likert rating scale. The questionnaire will provide information to assess glycemic control, and sub analysis of results related to diabetes management, problem solving and teaching. This scale ranges in score from 17 to 85, with higher scores consistent with increased self-efficacy.
Social Determinants of Health | 2 years
  The primary care giver will complete the 11-item "Health Leads USA Social Determinants of Health" questionnaire using a Yes/No rating scale to assess challenges with Social Determinants of Health
Caregiver Depression | 2 years
  The primary caregiver will complete the 9-item "Patient Health Questionnaire-9" using a 4-point Likert rating scale to assess their risk of depression. This scale ranges in score from 0 to 27, with higher scores consistent with increased risk of depression
Subject Depression | 2 years
  Subjects greater than 12 years old will complete the 13-item "Patient Health Questionnaire Modified for Adolescents" using a 4-point Likert rating scale and 4 Yes/No questions to assess their risk of depression. The Likert scale total ranges in score from 0 to 27, with higher scores consistent with increased risk of depression
Healthcare costs | 2 years
  Data will be extracted from the medical record of each patient to obtain information on healthcare charges and hospital reimbursement.

CONTACTS AND LOCATIONS:
Overall Officials: Colin P Hawkes, MD PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan K, Loar R, Anderson BJ, Heptulla RA. The role of socioeconomic status, depression, quality of life, and glycemic control in type 1 diabetes mellitus. J Pediatr. 2006 Oct;149(4):526-31. doi: 10.1016/j.jpeds.2006.05.039. PMID 17011326
- [Background] Kangovi S, Mitra N, Grande D, White ML, McCollum S, Sellman J, Shannon RP, Long JA. Patient-centered community health worker intervention to improve posthospital outcomes: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):535-43. doi: 10.1001/jamainternmed.2013.14327. PMID 24515422
- [Background] Raphael JL, Rueda A, Lion KC, Giordano TP. The role of lay health workers in pediatric chronic disease: a systematic review. Acad Pediatr. 2013 Sep-Oct;13(5):408-20. doi: 10.1016/j.acap.2013.04.015. PMID 24011745
- [Background] Katz ML, Volkening LK, Butler DA, Anderson BJ, Laffel LM. Family-based psychoeducation and Care Ambassador intervention to improve glycemic control in youth with type 1 diabetes: a randomized trial. Pediatr Diabetes. 2014 Mar;15(2):142-50. doi: 10.1111/pedi.12065. Epub 2013 Aug 5. PMID 23914987
- [Derived] Lai CW, Craven M, Hershey JA, Lipman TH, Hawkes CP. Adverse Social Determinants of Health in Children with Newly Diagnosed Type 1 Diabetes: A Potential Role for Community Health Workers. Pediatr Diabetes. 2024 Jan 23;2024:8810609. doi: 10.1155/2024/8810609. eCollection 2024. PMID 40302949